CLINICAL TRIAL: NCT00005832
Title: A Phase II Trial of R115777 (NSC #702818) in Patients With Advanced Pancreas Cancer
Brief Title: S9924 R115777 in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067846; S9924 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2004-04-26 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; duct cell adenocarcinoma of the pancreas; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R115777 (Experimental): 300mg/dose BID, PO, Days 1-21, q 28days
  Interventions: Drug: R115777

INTERVENTIONS:
Drug: R115777 — 300mg/dose BID, PO, Days 1-21, q 28days
  Other Names: tipifarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of R115777 in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the six month survival rate in patients with advanced adenocarcinoma of the pancreas treated with R115777. II. Determine the time to treatment failure and confirmed response in this patient population treated with this regimen. III. Evaluate the frequency and severity of toxicities associated with this treatment regimen in these patients.

OUTLINE: Patients receive oral R115777 twice daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed adenocarcinoma of the pancreas Ductal adenocarcinoma Mucinous noncystic carcinoma Signet ring cell carcinoma Adenosquamous carcinoma Undifferentiated (anaplastic) carcinoma Mixed ductal endocrine carcinoma Well differentiated adenocarcinoma Moderately well or poorly differentiated adenocarcinoma Undifferentiated ductal carcinoma No papillary cystic carcinomas, sarcomas, or tumors arising from the endocrine pancreas Pathological confirmation of a metastatic site allowed Clinical documentation of pancreatic involvement and no evidence of another primary allowed Locally advanced or distant metastatic disease surgically incurable No known brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Zubrod 0-1 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Ability to swallow and/or receive enteral medications via gastrostomy feeding tube No intractable nausea or vomiting No other prior malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer in remission Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent immunotherapy Chemotherapy: No prior chemotherapy No prior adjuvant or neoadjuvant chemoradiotherapy, including for advanced pancreatic cancer No other concurrent chemotherapy Endocrine therapy: No prior or concurrent hormonal therapy Radiotherapy: See Chemotherapy No prior radiotherapy, except for palliation to metastatic sites No concurrent radiotherapy Surgery: See Disease Characteristics At least 2 weeks since prior surgery for pancreatic cancer and recovered Prior partial resections of the stomach and duodenum for pancreatic cancer allowed No prior major resection of the small intestine Prior pancreaticduodenectomy for pancreatic cancer allowed Other: No concurrent proton pump inhibitors (e.g., omeprazole) Concurrent antacids or H2 blockers allowed No other concurrent therapy for pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2000-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Survival rate in patients with advanced adenocarcinoma of the pancreas treated with R115777 | 6 months

SECONDARY OUTCOMES:
Time to treatment failure | Once every 8 weeks until progression
Evaluate the frequency and severity of toxicities | Weekly for 8 weeks and then once every 4 weeks
Assess confirmed response (complete & partial) in patients with measurable advanced adenocarcinoma of the pancreas | Once every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S. MacDonald, MD, Study Chair — St. Vincent's Comprehensive Cancer Center - Manhattan
Locations (14):
- United States (14):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Macdonald JS, McCoy S, Whitehead RP, Iqbal S, Wade JL 3rd, Giguere JK, Abbruzzese JL. A phase II study of farnesyl transferase inhibitor R115777 in pancreatic cancer: a Southwest oncology group (SWOG 9924) study. Invest New Drugs. 2005 Oct;23(5):485-7. doi: 10.1007/s10637-005-2908-y. PMID 16133800
- [Result] Macdonald JS, Chansky K, Whitehead R, et al.: A phase II study of farnesyl transferase inhibitor R115777 in pancreatic cancer. A Southwest Oncology Group (SWOG) study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-548, 2002.